CLINICAL TRIAL: NCT03996863
Title: PUCE Study: Prevention of Unmitigated Chemotherapy-induced Emesis
Brief Title: Prevention of Unmitigated Chemotherapy-induced Emesis
Acronym: PUCE
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Drexel Oncology was shut down a few days before first patient in.
Sponsor: Otolith Labs (Industry)
Collaborators: Drexel University College of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: OLith10601
Record Dates: First submitted 2019-06-17; First posted 2019-06-25 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Chemotherapy-induced Nausea and Vomiting; Nausea Post Chemotherapy
Keywords: Nausea; Chemotherapy; cisplatin; Emesis
MeSH Terms: conditions — Vomiting; Nausea

STUDY DESIGN:
Intervention Model Description: Patients who qualify for the study based on their response to the first round of chemotherapy will be randomly assigned to one of two groups for their second and third rounds of chemotherapy.
  Half of the patients will be given a device set at working parameters believed to significantly mitigate nausea for their second round, and a placebo device for the third round of chemotherapy. The second half of the patients will receive the placebo device for the second round and the effective device for the third round.
Who Masked: Participant, Investigator
Masking Description: The sponsor will be randomly assigning the Otoband or placebo device to participants. The investigator will not know which device is assigned.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Otoband efficacy on CINV (Experimental): Participants will wear the Otoband during infusion following chemotherapy treatments, placed against the skin, on the flat part of the right mastoid bone.
  The Otoband will be able to function maximum 16 hours per day. Study participants will be instructed to use the device for 30 minutes in the morning, and then as needed for symptoms while at home for four days. Once the OtoBand is applied and turned on they are expected to wear it continually for up to 30 minutes. Subjects can stop the OtoBand 5 minutes after cessation of nausea but will be asked to resume stimulation if the nausea recurs within 30 minutes. The participant will be asked to fill out the MASCC Antiemesis Tool questionnaire at 24 hours post infusion and again at day 5 post infusion. Participants will also be asked to fill out an OtoBand Use Questionnaire daily for the four days following their chemotherapy infusion.
  Interventions: Device: Otoband
- Placebo device efficacy on CINV (Placebo Comparator): Participants will wear the placebo device during infusion following chemotherapy treatments, placed against the skin, on the flat part of the right mastoid bone.
  The placebo device will be able to function maximum 16 hours per day. Study participants will be instructed to use the device for 30 minutes in the morning, and then as needed for symptoms while at home for four days. Once the device is applied and turned on they are expected to wear it continually for up to 30 minutes. Subjects can stop the device 5 minutes after cessation of nausea but will be asked to resume stimulation if the nausea recurs within 30 minutes. The participant will be asked to fill out the MASCC Antiemesis Tool questionnaire at 24 hours post infusion and again at day 5 post infusion. Participants will also be asked to fill out an OtoBand Use Questionnaire daily for the four days following their chemotherapy infusion.
  Interventions: Device: Placebo device

INTERVENTIONS:
Device: Otoband — Participants during infusion following chemotherapy will wear the Otoband set at normal power (effective) for four days following treatment and nausea outcomes will be recorded by questionnaire or by the investigator during site visits.
  Arms: Otoband efficacy on CINV
Device: Placebo device — Participants during infusion following chemotherapy will wear the placebo device set at low power (6 decibels lower than normal power, ineffective power) for four days following treatment and nausea outcomes will be recorded by questionnaire or by the investigator during site visits.
  Arms: Placebo device efficacy on CINV

SUMMARY:
Chemotherapy-induced nausea and vomiting (CINV) remains a major obstacle to patient care and continues to decrease quality of life. Despite the addition of medications and antiemetic regimens, doctors' ability to control CINV is still inadequate: even moderately-emetogenic chemotherapy regimens cause roughly 20% of patients to have vomiting and over 40% to experience significant nausea. In this study, the investigators test a transcranial vibrating system that has shown great promise at reducing nausea and vomiting. .

DETAILED DESCRIPTION:
Chemotherapy-induced nausea and vomiting (CINV) remains a major obstacle to cancer patient care despite numerous medications being available to prevent and treat CINV.

CINV decreases quality of life in roughly one third of patients receiving highly emetogenic chemotherapy. In addition, roughly half to two thirds of all patients receiving chemotherapy require rescue anti-emetic medications despite being given guideline-based prophylactic anti-emetics.The anti-emesis armamentarium continues to grow with new medications, including olanzapine and fosaprepitant, being studied in recent years. However, despite the addition of these medications and guideline-based antiemetic regimens, the ability to control CINV is still inadequate as even moderately-emetogenic chemotherapy regimens cause roughly 20% of patients to have vomiting and over 40% to experience significant nausea.

In this study, the investigators aim to test a new transcranial vibrating system that has shown promise in phase I studies for treating dizziness, motion sickness and nausea.

ELIGIBILITY:
Inclusion Criteria:

* Subject currently receiving chemotherapy known to be emetogenic (i.e subject has already received one round of chemotherapy)
* MASCC Antiemesis Tool score of > 6 on the nausea severity scale and/or
* One or more episodes of vomiting anytime in the 4 days following receipt of chemotherapy and/or
* The need for three or more uses of rescue antiemetic medications within 4 days of chemotherapy during previous round.

Exclusion Criteria:

* Pregnant women
* Individuals unable to provide informed consent
* Any preexisting condition causing significant nausea or vomiting, or causing reaction to the bone conduction system (e.g. superior canal dehiscence)
* Prisoners

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
Change in MAT (MASCC Antiemesis Tool) score | MAT score is obtained on day 5 following each of the three chemotherapy treatments.
  Potential subjects will be screened for eligibility based on their responses to the (standard of care) questionnaire developed by the "Multinational Association for Supportive Care in Cancer" and called the MAT (Multinational Antiemesis Tool). MAT scores range from 0 (no issue) to 10 (most severe).
  Any difference in severity of nausea as measured by MAT score between active and placebo phases, and compared to the scores obtained in the pre-trial round of chemotherapy, will be analyzed.

SECONDARY OUTCOMES:
Change in number of episodes of vomiting | For the 5 days following each of the two chemotherapy infusions, with effective and placebo devices.
  The investigator will quantify any difference in the number of episodes of vomiting experienced because of chemotherapy-induced nausea and vomiting (CINV) between effective and placebo phases, and compare to the number of episodes that happened during the previous pre-trial chemotherapy session.
Change in amount of rescue antiemetics required to control chemotherapy-induced nausea and vomiting | For the 5 days following each of the two chemotherapy treatment.
  The investigator will quantify any difference in the amount of rescue antiemetics the patient chooses to control chemotherapy-induced nausea and vomiting (CINV) between effective and placebo phases, and compare to the amounts taken during the previous pre-trial chemotherapy session.
Change in population of "Complete responders" | For the 5 days following each of the two each chemotherapy treatment
  The investigator will quantify any difference in number of participants who are Complete Responders, as defined by a nausea severity scale on the MAT < 3, no vomiting, and no use of rescue antiemetics for the complete 4 days following chemotherapy infusion, between acute and placebo phases.

CONTACTS AND LOCATIONS:
Overall Officials: Michael S Sherman, MD, Principal Investigator — Drexel University College of Medicine
Locations (1):
- I. Brodsky Associates Outpatient Hematology & Oncology Clinic, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kottschade L, Novotny P, Lyss A, Mazurczak M, Loprinzi C, Barton D. Chemotherapy-induced nausea and vomiting: incidence and characteristics of persistent symptoms and future directions NCCTG N08C3 (Alliance). Support Care Cancer. 2016 Jun;24(6):2661-7. doi: 10.1007/s00520-016-3080-y. Epub 2016 Jan 15. PMID 26768436
- [Background] Lindley CM, Bernard S, Fields SM. Incidence and duration of chemotherapy-induced nausea and vomiting in the outpatient oncology population. J Clin Oncol. 1989 Aug;7(8):1142-9. doi: 10.1200/JCO.1989.7.8.1142. PMID 2787840
- [Background] Escobar Y, Cajaraville G, Virizuela JA, Alvarez R, Munoz A, Olariaga O, Tames MJ, Muros B, Lecumberri MJ, Feliu J, Martinez P, Adansa JC, Martinez MJ, Lopez R, Blasco A, Gascon P, Calvo V, Luna P, Montalar J, Del Barrio P, Tornamira MV. Incidence of chemotherapy-induced nausea and vomiting with moderately emetogenic chemotherapy: ADVICE (Actual Data of Vomiting Incidence by Chemotherapy Evaluation) study. Support Care Cancer. 2015 Sep;23(9):2833-40. doi: 10.1007/s00520-015-2809-3. Epub 2015 Jun 17. PMID 26081597